CLINICAL TRIAL: NCT06974162
Title: Metagenomic Sequencing of Ocular Fluids in Patients With Ocular Inflammation
Brief Title: Metagenomics for Ocular Inflammation
Status: Recruiting | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CHUC1004; 25/WM/0072 (Other: NHS Health Research Authority); 354543 (Other: IRAS Project ID)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Uveitis; Aqueous Humor; Infection
Keywords: Metagenomics; Uveitis; Aqueous Humor; Ophthalmology
MeSH Terms: conditions — Uveitis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metagenomic Sequencing on aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ocular inflammation presumed to be infectious or para-infectious: Patients with Ocular Inflammation undergoing Metagenomics on Aqueous Humour
  Interventions: Diagnostic Test: Metagenomic sequencing of aqueous humor; Diagnostic Test: Ocular Imaging

INTERVENTIONS:
Diagnostic Test: Metagenomic sequencing of aqueous humor — Metagenomic Sequencing on aqueous humor surplus to diagnostic requirements
Diagnostic Test: Ocular Imaging — Ocular imaging with anterior segment OCT, laser flare photometry, confocal microscopy and colour fundus photography.

SUMMARY:
The aim of this study is to apply a diagnostic test called 'metagenomic sequencing' to identify the involvement of potential infections in patients with ocular inflammation, where this hasn't been detected by currently available standard testing. For many people with ocular inflammation, no cause is ever found for their disease. In some cases, an infection or infectious trigger is suspected, but currently available tests are inadequate. Metagenomic sequencing can identify almost every globally known infection (bacteria, virus, fungi, parasites) in a sample. Therefore, it has the potential to identify an infection that has caused or triggered ocular inflammation, and as a consequence may help to identify specific treatments. It has the potential to improve our understanding of how to diagnose and treat people with this problem. This study will allow us to test the technique that has been previously optimised for brain infections, on ocular fluids. Participants will be 18 years of age or over and have active ocular inflammation which is suspected to be due to an infection, or an autoimmune process which has been triggered by an infection, but identification of this infection has not been possible using the investigations available as part of standard NHS care. Participants will be identified by the treating clinical team as requiring a sample of fluid from inside of the eye, and some of this fluid will be sent for metagenomic sequencing alongside standard testing. This study will be conducted at Moorfields Eye Hospital, London and will last for approximately a year. Participants will undergo additional non-invasive ocular imaging on the day of their clinic visit, but will not have to attend any additional research visits.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older with the capacity to consent
2. Standard of care has not determined a clinical diagnosis
3. Active ocular inflammation with risk of visual loss
4. Clinically suspected infectious or para-infectious cause of ocular inflammation

Exclusion Criteria:

1. Contraindication to ocular fluid sampling
2. Where an urgent result within 5 days is clinically required

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the UK attending Moorfields Eye Hospital, London.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants who receive a clinically viable result from metagenomic sequencing | 12 months

SECONDARY OUTCOMES:
The number of patients who receive a result that leads to a change in treatment and beneficial outcome from metagenomic sequencing | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant demographics and research findings will be shared in the peer-reviewed scientific publication.
Supporting Information: Study Protocol
Time Frame: Within 12 months of study completion, for 5 years held in the Clinical Research Facility at Moorfields Eye Hospital.
Access Criteria: On request to Moorfields Eye Hospital
URL: https://www.moorfields.nhs.uk/research/nihr-moorfields-clinical-research-facility-crf

REFERENCES:
- [Background] Atkinson L, Lee JC, Lennon A, Shah D, Storey N, Morfopoulou S, Harris KA, Breuer J, Brown JR. Untargeted metagenomics protocol for the diagnosis of infection from CSF and tissue from sterile sites. Heliyon. 2023 Sep 9;9(9):e19854. doi: 10.1016/j.heliyon.2023.e19854. eCollection 2023 Sep. PMID 37809666
- [Background] Penner J, Hassell J, Brown JR, Mankad K, Storey N, Atkinson L, Ranganathan N, Lennon A, Lee JCD, Champsas D, Kopec A, Shah D, Venturini C, Dixon G, De S, Hatcher J, Harris K, Aquilina K, Kusters MA, Moshal K, Shingadia D, Worth AJJ, Lucchini G, Merve A, Jacques TS, Bamford A, Kaliakatsos M, Breuer J, Morfopoulou S. Translating metagenomics into clinical practice for complex paediatric neurological presentations. J Infect. 2023 Nov;87(5):451-458. doi: 10.1016/j.jinf.2023.08.002. Epub 2023 Aug 7. No abstract available. PMID 37557958
- [Background] Doan T, Acharya NR, Pinsky BA, Sahoo MK, Chow ED, Banaei N, Budvytiene I, Cevallos V, Zhong L, Zhou Z, Lietman TM, DeRisi JL. Metagenomic DNA Sequencing for the Diagnosis of Intraocular Infections. Ophthalmology. 2017 Aug;124(8):1247-1248. doi: 10.1016/j.ophtha.2017.03.045. Epub 2017 May 16. No abstract available. PMID 28526549
- See also: Related Info — https://www.moorfields.nhs.uk/research/nihr-moorfields-clinical-research-facility-crf